CLINICAL TRIAL: NCT04153981
Title: A Multicenter, Open-Label, Single-Arm, Phase 4 Study to Assess the Safety of Basaglar in Subjects With Type 2 Diabetes Mellitus in India
Brief Title: A Study of Insulin Glargine (LY2963016) in Adult Participants With Type 2 Diabetes in India
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17225; I4L-IN-ABEX (Other: Eli Lilly and Company)
Record Dates: First submitted 2019-11-05; First posted 2019-11-06 (Actual); Results first posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; LY2963016 insulin glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insulin Glargine (Experimental): Participants received insulin glargine once a day (QD) subcutaneously (SC) with a starting dose of 10 units. Participants self-titrated once or twice weekly until fasting blood glucose level was lowered to <100 milligrams per deciliter (mg/dL). Dose was reduced by 4 units in case of hypoglycemia.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Glargine — Administered SC
  Other Names: LY2963016; Basaglar

SUMMARY:
The reason for this study is to see if insulin glargine is safe in participants with type 2 diabetes mellitus (T2DM) in India.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM based on the disease diagnostic criteria from the World Health Organization (WHO) classification for at least 6 months before screening.
* Have been receiving glucagon-like peptide-1 receptor agonist (GLP-1 RA) or ≥2 oral antihyperglycemic medication (OAMs) at stable doses for 90 days prior to screening.
* Have an HbA1c level ≥7.0% and <11.0%.
* Have never been treated with insulins except for short term treatment of acute conditions up to a maximum of 14 days.

Exclusion Criteria:

* Have any form of diabetes other than T2DM.
* Have hypersensitivity to the active substance of LY2963016 or to any of the excipients.
* Have any clinically significant disorder, other than T2DM, that in the investigator's opinion, would preclude participation in the trial.
* Are receiving systemic glucocorticosteroids therapy or have excessive insulin resistance (total insulin dose >2 units per kilogram).
* Have a history or diagnosis of human immunodeficiency virus infection, hepatitis B and C.
* Have comorbidities of unstable angina, cardiac failure (Stage III or IV as per New York Heart Association guidelines) or renal failure (estimated glomerular filtration rate <30 milliliters/minute/meter squared).
* Are pregnant or intend to become pregnant during the course of the study; or are sexually active women of child-bearing potential not actively practicing birth control by a medically acceptable method as determined by the investigator.
* Is a woman who is breastfeeding.
* Have participated within the last 30 days in a clinical trial involving an investigational product other than the LY2963016. If the previous investigational product has a long half-life, 3 months or 5 half-lives (whichever is longer) should have passed.
* Have previously completed or withdrawn from this study or any other study investigating LY2963016. This exclusion criterion does not apply to participants who are rescreened prior to baseline visit.
* Are currently enrolled in any other clinical study involving an investigational product or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Are unwilling or unable to comply with the use of a glucometer.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (11):
- India (11):
  - DIACARE, Ahemdabad, Gujarat
  - Gujarat Endocrine Center, Ahmedabad, Gujarat
  - Nirmal Hospital Private Limited, Surat, Gujarat
  - Government Medical College & Sir Sayajirao General Hospital, Vadodara, Gujarat
  - Sumandeep Vidhyapeeth & Dhiraj General Hospital, Vadodara, Gujarat
  - Bangalore Diabetes Center, Bangalore, Karnataka
  - Supe Heart & Diabetes Hospital & Research Centre, Nashik, Maharashtra
  - Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi
  - GSVM Medical College, Kanpur, Uttar Pradesh
  - Popular Hospital, Varanasi, Uttar Pradesh
  - Maharaja Agrasen Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Insulin Glargine
Started | 304
Participants Who Received At Least One Dose of Study Drug | 259
Completed | 218
Not Completed | 86
Not completed — Death | 1
Not completed — Withdrawal by Subject | 24
Not completed — Lost to Follow-up | 1
Not completed — Physician Decision | 1
Not completed — Due to Unavailable Glucometer | 1
Not completed — Covid 19 | 52
Not completed — Participant Dropped Out as Required Laboratory Test was Not Performed | 5
Not completed — Due to Low Fasting Blood Sugar Levels | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Insulin Glargine: Participants received insulin glargine QD SC with a starting dose of 10 units. Participants self-titrated once or twice weekly until fasting blood glucose level was lowered to <100 mg/dL. Dose was reduced by 4 units in case of hypoglycemia.
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 259
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.1 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93
  Male | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 259
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  India | 259

OUTCOME MEASURES:

1. Primary Outcome: Number or Participants With Hypoglycemic Events
Description: Hypoglycemic event is when the fasting blood glucose (FBG) level is ≤ 54 milligrams per deciliter (mg/dL) [≤ 3.0 millimoles per liter (mmol/L)].
Time Frame: Baseline to Week 24
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 259
participants | 10

2. Secondary Outcome: Basal Insulin Dose
Description: Basal Insulin Dose at Week 24.
Time Frame: Week 24
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: Units per kilograms per day (U/kg/day)
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 259
Units per kilograms per day (U/kg/day) | 0.30 (0.116)

3. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight was evaluated. Least Square (LS) mean was calculated using generalized linear model with the analysis variable as outcome, and the baseline of the analysis variable as covariate.
Time Frame: Baseline, Week 24
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 259
kilogram (kg) | -0.5 (0.15)

4. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: HbA1c is the glycosylated fraction of hemoglobin A. HbA1c is measured to identify average plasma glucose concentration over prolonged periods of time. LS mean was calculated using generalized linear model with the analysis variable as outcome, and the baseline of analysis variable as covariate.
Time Frame: Baseline, Week 12 and Week 24
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 259
Percentage of HbA1c
  At Week 12 | -0.641 (0.0719)
  At Week 24 | -0.860 (0.0847)

5. Secondary Outcome: Change From Baseline in 7-Point Self-Monitoring Blood Glucose (SMBG) Values
Description: Seven-point SMBG was completed at the following timepoints: Before Breakfast, 2 Hours After Morning Meal, Before Mid-Day Meal, 2 Hours After Mid-Day Meal, Before Evening Meal, 2 Hours After Evening Meal and at 3 AM (± 1 hour). LS mean was calculated using generalized linear model with the analysis variable as outcome, and the baseline of analysis variable as covariate.
Time Frame: Baseline, Week 24
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: milligrams per deciliter (mg/dL)
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 259
milligrams per deciliter (mg/dL)
  Blood glucose concentration before breakfast | -38.7 (2.12)
  Blood glucose concentration 2 hours after morning meal | -54.3 (2.87)
  Blood glucose concentration before midday meal | -32.9 (2.52)
  Blood glucose concentration 2 hours after midday meal | -43.6 (2.98)
  Blood glucose concentration before evening meal | -29.4 (2.41)
  Blood glucose concentration 2 hours after evening meal | -45.7 (2.97)
  Blood glucose concentration at 3AM (± 1 hour) | -32.9 (2.20)

6. Secondary Outcome: Change From Week 4 in Insulin Treatment Satisfaction Questionnaire (ITSQ)
Description: The ITSQ is a 22-item questionnaire that assesses treatment satisfaction for participants taking insulin, under 5 domains: Inconvenience of Regimen [(IR) - 5 items], Lifestyle Flexibility [(LF) - 3 items], Glycemic Control [(GC) - 3 items], Hypoglycemic Control [(HC) - 5 items], Insulin Delivery Device [(IDD) - 6 items]. Each Item is measured on a 7-point scale, with scores ranging for IR from 5 to 35, LF from 3 to 21, GC from 3 to 21, HC from 5 to 35, IDD from 6 to 42. Lower scores reflect better outcomes. LS mean was calculated using generalized linear model with the analysis variable as outcome, and the baseline of analysis variable as covariate. ITSQ was not evaluated at Week 0. For this outcome, Week 4 was considered as baseline.
Time Frame: Baseline (Week 4), Week 24
Population: All participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Insulin Glargine
Number analyzed (Participants) | 259
score on a scale
  ITSQ IR Score | -0.3 (0.04)
  ITSQ LF Score | -0.3 (0.05)
  ITSQ GC Score | -0.2 (0.05)
  ITSQ HC Score | -0.3 (0.05)
  ITSQ IDD Score | -0.3 (0.04)

ADVERSE EVENTS:
Time Frame: Up to 28 weeks
Description: All participants who received at least one dose of study drug.
Arm/Group | Insulin Glargine
All-Cause Mortality (participants affected / at risk) | 1/259
Serious Adverse Events (participants affected / at risk) | 1/259
Other Adverse Events (participants affected / at risk) | 8/259
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine (N=259)
Death (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine (N=259)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Pyrexia (General disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-10-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT04153981/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/81/NCT04153981/SAP_001.pdf